CLINICAL TRIAL: NCT01503944
Title: Detection of Striatal Dopaminergic Degeneration and Neocortical Amyloid Pathology in Patients With Dementia With Lewy Bodies, Alzheimer's Disease, Parkinson's Disease, and Healthy Elderly Volunteers
Brief Title: A Trial of 18F-AV-133 and 18F-AV-45 Positron Emission Tomography (PET)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-133-B03
Record Dates: First submitted 2010-07-14; First posted 2012-01-04 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Dementia With Lewy Bodies; Alzheimer's Disease; Parkinson's Disease
MeSH Terms: conditions — Lewy Body Disease; Alzheimer Disease; Parkinson Disease | interventions — florbenazine F 18; florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dementia with Lewy Bodies (Other)
  Interventions: Drug: 18F-AV-133; Drug: 18F-AV-45
- Parkinson's disease (Other)
  Interventions: Drug: 18F-AV-133; Drug: 18F-AV-45
- Healthy Elderly Volunteers (Other)
  Interventions: Drug: 18F-AV-133; Drug: 18F-AV-45
- Alzheimer's Disease (Other)
  Interventions: Drug: 18F-AV-133; Drug: 18F-AV-45

INTERVENTIONS:
Drug: 18F-AV-133 — 185 MBq
Drug: 18F-AV-45 — 185-370 MBq

SUMMARY:
The purpose of this study is to evaluate the ability to identify individuals with dopaminergic degeneration in group of patients with a clinical diagnosis of either dementia with Lewy bodies (DLB) or idiopathic Parkinson's disease and to differentiate them from Alzheimer's disease (AD) and control subjects.

ELIGIBILITY:
Inclusion Criteria DLB:

* Male or female > 50 years of age
* Meet the diagnostic criteria for probable DLB as established by the DLB Consortium (McKeith et al., 2005)

Inclusion Criteria AD:

* Male or female > 50 years of age
* Meet the NINCDS criteria for probable AD and have a Mini Mental State Examination (MMSE) score at screening between 10 and 24 inclusive

Inclusion Criteria PD:

* Male or female > 50 years of age
* Have probable PD according to the following criteria (Gelb et al., 1999):

  * Presence of 2 of the following 3 features: rest tremor, rigidity, bradykinesia;
  * Documented history of a sustained (>6 months) improvement to Levodopa (L-DOPA) or a dopamine agonist
  * Absence of atypical clinical features or other possible signs or symptoms suggesting another cause of parkinsonism such as a history of frequent falls as a prominent early feature, localized brain lesion(s) or neuroleptic use
  * Asymmetric onset
* A diagnosis of PD made within the 4 years prior to enrollment

Normal subjects:

* Are males or females > 50 years of age
* Have a MMSE score > 29, and are cognitively normal on the psychometric test battery at screening
* Have no signs or symptoms of clinically meaningful parkinsonism

Exclusion Criteria:

* Have a history or current diagnosis of other neurologic disease
* Have evidence of clinically significant cerebrovascular disease
* Have evidence from MRI or other biomarker studies that suggests the presence of a CNS pathology other than that associated with the study diseases

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
18F-AV-133 striatal to occipital standard uptake value ratio | Four Weeks
  The ratio of tracer activity in striatal target areas of interest relative to the occipital cortex reference region

SECONDARY OUTCOMES:
18F-AV-45 cortical to cerebellar standard uptake value ratio | Four Weeks
  The ratio of tracer activity in cortical target areas of interest relative to the cerebellum reference region

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (2):
- United States (2):
  - Research Site, Sun City, Arizona
  - Research Site, Philadelphia, Pennsylvania